CLINICAL TRIAL: NCT05069883
Title: Role of Oral Steroids in Reducing Recurrence of Urethral Stricture After Direct Vision Internal Urethrotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Collaborators: Armed Forces Institute of Urology, Rawalpindi (Other)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principal Investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AF1
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-03

CONDITIONS: Recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Steroid (Experimental): In this group oral steroids were given after Direct vision internal urethrotomy
  Interventions: Drug: Steroid Drug
- No Oral Steroids (Placebo Comparator): In this group no oral steroids were given after Direct vision internal urethrotomy
  Interventions: Drug: No steroid

INTERVENTIONS:
Drug: Steroid Drug — In this group Oral steroid medication after Direct Vision Internal Urethrotomy
  Other Names: Oral steroid medication
  Arms: Oral Steroid
Drug: No steroid — In this group no Oral steroid medication (palcebo medication) after Direct Vision Internal Urethrotomy
  Other Names: Placebo Medication
  Arms: No Oral Steroids

SUMMARY:
It was a randomized controlled trial conducted at department of Urology, Armed Forces Institute of Urology, Rawalpindi from 1st January, 2018 July 2019 to 31st March 2021 to determine the role of oral steroids after Direct Vision Internal Urethrotomy to reduce the recurrence rate of urethral strictures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urethral stricture with restricted urine flow of < 15 ml/min on uroflowmetry

Exclusion Criteria:

* Patients presenting with post-anastomotic urethroplasty strictures (assessed on history and medical record),
* Patients with post-TURP strictures
* Patients with neurogenic bladder
* Patients with prior history of steroid use
* Patients with extravasation during optical internal urethrotomy

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Recurrence of Urethral Stricture | 6 months post-operatively
  Number of patients presenting with recurrence of urethral stricture after direct vision internal urethrotomy

CONTACTS AND LOCATIONS:
Overall Officials: Barza Afzal, MBBS, FCPS, Study Director — barza_afzal@hotmail.com
Locations (1):
- Armed Force Institute of Urology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided